CLINICAL TRIAL: NCT03161028
Title: Lipoic Acid for the Treatment of Progressive Multiple Sclerosis
Brief Title: Lipoic Acid for Progressive Multiple Sclerosis (MS)
Acronym: LAPMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2682-R
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; magnetic resonance imaging; gait; neuroprotective agents; thioctic acid; alpha-lipoic acid; mobility; chronic progressive multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Lipoic Acid (Experimental): 59 subjects receive oral lipoic acid 1200mg daily
  Interventions: Drug: Lipoic acid
- Arm 2: Placebo (Placebo Comparator): 59 subjects receive placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lipoic acid — 1200 mg taken by mouth daily for two years starting on day one of the study and ending on the last day of study participation.
  Other Names: Alpha-lipoic acid
  Arms: Arm 1: Lipoic Acid
Drug: Placebo — The placebo comparator will be taken by mouth daily for two years starting on day one of the study and ending on the last day of study participation
  Arms: Arm 2: Placebo

SUMMARY:
The purpose of the study is to determine if lipoic acid can preserve mobility and protect the brain in progressive forms of multiple sclerosis.

DETAILED DESCRIPTION:
This two-year study will determine if daily oral intake of lipoic acid will prove superior to placebo in reducing injury to the brain and maintaining mobility in progressive MS. Mobility will be assessed with the timed 25-foot walk test and 2-minute timed walk test as well as fall counts. Neuroprotection will be measured by the extent of brain volume loss seen on MRI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of progressive MS as defined by the study
* Able to give informed consent and to adhere to study procedures.
* Expanded Disability Status Scale (EDSS) 3.0 - 6.5: ambulatory for at least 20 meters without rest and use of bilateral aids (canes, crutches, walker) or better.

Exclusion Criteria:

* A self-reported medical or neurological problem other than MS that is a cause of progressive or fluctuating gait dysfunction
* Unable to undergo MRI
* Unable to follow directions in English as standardized scales are not all validated in other languages.
* Current major disease or disorder other than MS (e.g., cancer, renal disease, end-stage cardiopulmonary disease, post-traumatic stress disorder, etc.) that may interfere with study procedures. Note: Stable abnormal laboratory values of no more than Grade 1 determined to not be of clinical significance to the primary treating physician for that condition may be permitted per local site investigator discretion.
* Pregnant or breast-feeding.
* Insulin-dependent diabetes or diabetes not controlled on oral diabetes medications.
* Scheduled (every 3 months or more frequently) IV or oral steroids in the year prior to enrolment.
* IV or oral steroids in the 60 days prior to enrolment.
* Use of LA in the prior 2 years exceeding the equivalent of 1200mg daily for 3 months.
* Participation in the pilot LA in SPMS trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca I. Spain, MD MSPH, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (11):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Colorado, Aurora, Colorado
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spain RI, Paz Soldan MM, Freedman MS, Repovic P, Solomon AJ, Rinker JR, Wallin MT, Haselkorn JK, Stuve O, Gross RH, Waslo CS, Hildebrand A, Morris CD, Mitchell J, Turner AP, Schwartz DL, Metz J, Rooney W. Lipoic Acid for Treatment of Progressive Multiple Sclerosis: A Phase 2 Randomized Clinical Trial. Neurology. 2026 Jan 13;106(1):e214454. doi: 10.1212/WNL.0000000000214454. Epub 2025 Dec 15. PMID 41397213
- [Derived] Spain RI, Hildebrand A, Waslo CS, Rooney WD, Emmons J, Schwartz DL, Freedman MS, Paz Soldan MM, Repovic P, Solomon AJ, Rinker J 2nd, Wallin M, Haselkorn JK, Stuve O, Gross RH, Turner AP. Processing speed and memory test performance are associated with different brain region volumes in Veterans and others with progressive multiple sclerosis. Front Neurol. 2023 Jun 8;14:1188124. doi: 10.3389/fneur.2023.1188124. eCollection 2023. PMID 37360346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 Veteran Affairs Medical Centers, 1 Medical Health System, and 5 US and Canada University Hospitals. The first participant was enrolled on August 17, 2018 and the last participant was enrolled in January 2022.
Groups:
- Lipoic Acid: Participants received 1200mg daily lipoic acid orally for 24 months. Lipoic acid: 1200 mg capsule
- Placebo: Participants received placebo capsule matching lipoic acid orally for 24 months.
  Placebo: lipoic acid placebo capsule
Period: Overall Study
Arm/Group | Lipoic Acid | Placebo
Started | 54 | 61
Completed | 34 | 51
Not Completed | 20 | 10
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Adverse Event | 5 | 1
Not completed — Study drug side effects | 2 | 2
Not completed — Administrative PD/UP | 4 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Unable to comply with procedures | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lipoic Acid | Placebo | Total
Number analyzed (Participants) | 54 | 61 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.5) | 58.6 (7.7) | 59.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 25 | 27 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 50 | 55 | 105
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 8 | 7 | 15
  United States | 46 | 54 | 100
MS Subtype [Count of Participants; unit: Participants]
  Primary progressive MS (PPMS) | 16 | 18 | 34
  Secondary progressive MS (SPMS) | 38 | 43 | 81
EDSS [Median (Inter-Quartile Range); unit: score] — Expanded Disability Status Scale (EDSS) is a tool used to measure the level of disability in people with MS. Scale ranges from 0 to 10, with higher scores indicating greater disability.
  score | 6.0 [4.0 to 6.5] | 6.0 [4.0 to 6.0] | 6.0 [4.0 to 6.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Mobility: Timed 25 Foot Walk
Description: T25FW was transformed to walking speed by dividing 25 feet by the completion time in seconds (ft/sec). The change in walking speed across 24 months was compared between treatment groups using a mixed models analysis.
Time Frame: 24 months
Population: Intent to Treat Population (all participants assigned to lipoic acid or placebo).
Measure: Mean (95% Confidence Interval); unit: feet per second
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 54 | 61
feet per second | -0.39 [-0.58 to -0.20] | -0.30 [-0.46 to -0.14]
Statistical Analysis 1: Comparison: Lipoic Acid vs Placebo; For the model evaluating the primary outcome (change in T25FW), T25FW was transformed to walking speed by dividing 25 feet by the completion time in seconds (ft/sec). Any participants who were unable to complete the T25FW at any timepoint after baseline were assigned a value of 199 seconds, a statistical technique known as Winsorizing; Test type: Superiority; p = 0.51, Mixed Models Analysis — The threshold for statistical significance was p = 0.05

2. Secondary Outcome: Change in Mobility: 2-minute Timed Walk
Description: The score is the distance, in meters, the subject walks in 2 minutes. The change in walking distance across 24 months was compared between treatment groups using a mixed models analysis.
Time Frame: 24 months
Population: Intent to Treat Population (all participants assigned to lipoic acid or placebo).
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 54 | 61
meters | -7.25 [-16.57 to 2.07] | -8.02 [-15.97 to -0.08]
Statistical Analysis 1: Comparison: Lipoic Acid vs Placebo; Test type: Superiority; p = 0.902, Mixed Models Analysis

3. Secondary Outcome: Mobility: Fall Count
Description: Change in number of falls recorded from Baseline to year 2
Time Frame: 24 months
Population: Intent to Treat Population (all participants assigned to lipoic acid or placebo).
Measure: Mean (Inter-Quartile Range); unit: Falls
Groups:
- Arm 1: Lipoic Acid: 54 subjects receive oral lipoic acid 1200mg daily
  Lipoic acid: 1200 mg taken by mouth daily for two years starting on day one of the study and ending on the last day of study participation.
- Arm 2: Placebo: 61 subjects receive placebo daily
  Placebo: The placebo comparator will be taken by mouth daily for two years starting on day one of the study and ending on the last day of study participation
Arm/Group | Arm 1: Lipoic Acid | Arm 2: Placebo
Number analyzed (Participants) | 54 | 61
Falls | 0.65 [0.30 to 1.39] | 0.63 [0.33 to 1.18]
Statistical Analysis 1: Comparison: Arm 1: Lipoic Acid vs Arm 2: Placebo; Test type: Superiority; p = 0.90, Mixed Models Analysis

4. Secondary Outcome: Brain Atrophy by MRI
Description: Change in whole brain volume from baseline to 24 months
Time Frame: 24 months
Population: Intent to Treat Population (all participants assigned to lipoic acid or placebo).
Measure: Mean (95% Confidence Interval); unit: cm3
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 54 | 61
cm3 | -0.58 [-6.29 to 5.13] | -7.18 [-11.95 to -2.40]
Statistical Analysis 1: Comparison: Lipoic Acid vs Placebo; Test type: Superiority; p = 0.084, Mixed Models Analysis

5. Other Pre Specified Outcome: Safety: Adverse Event Monitoring
Description: Participants with at least 1 treatment-emergent AE
Time Frame: 24 months
Population: Intent to Treat Population (all participants assigned to lipoic acid or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 54 | 61
Participants | 35 | 30
Statistical Analysis 1: Comparison: Lipoic Acid vs Placebo; Test type: Superiority; p = 0.134, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 years of treatment
Description: AE and laboratory abnormalities were captured and categorized using the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). The Suicide Behaviors Questionnaire-Revised (SBQ-R) was used to monitor for suicidality as required by the Food & Drug Administration.
Arm/Group | Lipoic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/54 | 1/61
Serious Adverse Events (participants affected / at risk) | 11/54 | 7/61
Other Adverse Events (participants affected / at risk) | 35/54 | 30/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipoic Acid (N=54) | Placebo (N=61)
Clostridium difficile colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute hypoxic hypercarbic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Vascular disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chest pain (non-cardiac) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cholecystitis NOS (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Injurious fall
Muscular weakness (Nervous system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pelvic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Traumatic haemothorax (Vascular disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pneumonia NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 2 (2)
Syncope (Vascular disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipoic Acid (N=54) | Placebo (N=61)
Glomerular filtration rate decreased (Investigations) | 13 (15) | 9 (12)
Proteinuria (Renal and urinary disorders) | 11 (14) | 2 (2)
Alanine aminotransferase increased (Investigations) | 6 (6) | 8 (9)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 3 (4)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 9 (14)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitations of the study include issues of low power, COVID-19 pandemic interruptions in study recruitment and data collection, and unexpected study withdrawals due to proteinuria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT03161028/Prot_SAP_000.pdf